CLINICAL TRIAL: NCT07257900
Title: Effects of Video Game-Based Exercise Training on Physical Activity, Balance, Fatigue, and Quality of Life in Pediatric-Onset Multiple Sclerosis Patients
Brief Title: Comparison of Structured Exercise and Exergaming in Pediatric-Onset Multiple Sclerosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Melisa Topaloglu, Physiotherapist, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IUC-POMS-EXERGAME-2025
Record Dates: First submitted 2025-11-17; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Pediatric-Onset Multiple Sclerosis (POMS); Exercise Training
Keywords: Pediatric-onset multiple sclerosis; Physiotherapy; Exergaming; Exercises; telerehabilitation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured Functional Exercise Training (Experimental): Participants in this group will receive a supervised, home-based physiotherapy program delivered via Zoom, including aerobic, strengthening, balance, and coordination exercises. Sessions will take place twice per week for 8 weeks, 45-60 minutes each.
  Interventions: Behavioral: Structured Functional Exercise Program
- Exergaming-Based Rehabilitation (Experimental): Participants in this group will perform interactive motion-based games designed to improve physical activity, strength, balance, and motivation. The exergaming sessions will be held twice per week for 8 weeks, each lasting 45-60 minutes, supervised by a physiotherapist.
  Interventions: Behavioral: Exergaming Rehabilitation

INTERVENTIONS:
Behavioral: Structured Functional Exercise Program — Sessions will be conducted twice per week for 8 weeks via live online video conferencing (Zoom) under the supervision of a physiotherapist. Each session will last 45-60 minutes and include aerobic, strengthening, and balance exercises adapted for home environments. At the beginning of the program, there will be approximately 5 minutes of low-to-moderate intensity warm-up exercises, followed by approximately 20 minutes of aerobic exercises, approximately 20 minutes of strength and balance exercises, and 5 minutes of cool-down exercises. These exercises are structured with increasing intensity over the weeks.
  * Weeks 1-2: 2 sets x 10 reps
  * Weeks 3-4: 2 sets x 15 reps
  * Weeks 5-6: 2 sets x 10 reps, with half a kilo added for the upper extremities and one kilo added for the lower extremities.
  * Weeks 7-8: 2 sets x 15 reps with free weights
  Arms: Structured Functional Exercise Training
Behavioral: Exergaming Rehabilitation — The intervention will use interactive motion-based video games, such as the Nintendo Switch Ring Fit Adventure™ platform, incorporating aerobic, strengthening, and balance activities. Each session will provide visual and auditory feedback to promote motivation and adherence. Sessions will be conducted twice per week for 8 weeks under physiotherapist supervision.It will be implemented at three levels: beginner, intermediate, and advanced. The number of repetitions and difficulty levels will be gradually increased. The first two weeks will be at the beginner level, weeks 3-5 at the intermediate level, and weeks 6-8 at the advanced level. The session will begin with a 5-minute warm-up, followed by approximately 20 minutes of aerobic exercises, approximately 20 minutes of strength and balance exercises, and conclude with a 5-minute cool-down. The program's exergame training activities include jogging, mini games, strength training, balance, and yoga exercises.
  Arms: Exergaming-Based Rehabilitation

SUMMARY:
This study will examine how two different exercise programs affect children and young adults with pediatric-onset multiple sclerosis (POMS). POMS is a type of multiple sclerosis that begins in childhood or adolescence and can cause fatigue, weakness, balance problems, and difficulty moving. This study aims to evaluate the effectiveness of a video game-based exercise program (exergaming) compared with traditional exercise training in enhancing balance, physical activity levels, reducing fatigue, and improving quality of life in individuals with pediatric-onset multiple sclerosis. Approximately 30 participants aged 12 to 22 years old who have been diagnosed with POMS and have mild to moderate symptoms (Extended Disability Status Scale [EDSS] score below 6) will participate in the study.

Participants will be randomly assigned to one of two groups:

Traditional Exercise Group: Participants will receive structured exercise instruction via live Zoom sessions (a tele-rehabilitation model). For 8 weeks, twice a week, they will perform supervised aerobic, strength, and balance exercises, each lasting approximately 45 minutes.

Exercise Game Group: Participants will perform similar aerobic, strength training, and balance exercises using the Nintendo Switch Ring Fit Adventure™ video game system.

Researchers will evaluate participants' physical activity levels, balance, fatigue, and quality of life parameters at baseline and after completing the 8-week intervention.

The study aims to determine whether the exergaming program can help participants increase their physical activity, reduce fatigue, and improve balance and daily functioning compared with traditional exercise. This approach offers an engaging and technology-supported way to incorporate physical activity into the rehabilitation of young people with POMS.

DETAILED DESCRIPTION:
Pediatric-onset multiple sclerosis (POMS) is a chronic demyelinating disorder of the central nervous system that begins in childhood or adolescence. It causes lifelong physical and cognitive limitations. Individuals with POMS often experience decreased motor abilities, balance impairments, and fatigue. These symptoms can lower quality of life (Chitnis et al., 2009; Prajjwal et al., 2023). Regular exercise plays a vital role in preserving and improving physical capacity in individuals with multiple sclerosis. However, maintaining adherence to exercise programs among children and adolescents remains a major challenge. Studies have shown that pediatric MS patients often find traditional physiotherapy programs monotonous and may avoid exercise due to fatigue or fear of relapse (Sikes et al., 2019). Exergaming, defined as video game-based physical activity, has emerged as a promising rehabilitation tool. It combines physical exercise with motivational and interactive game elements. By providing real-time feedback, sensory engagement, and enjoyment, exergaming may increase adherence and participation in rehabilitation programs. Previous research has reported positive effects of exergaming on balance, fatigue, and quality of life in various neurological populations (Motl & Pilutti, 2016; Polizzi et al., 2024). However, there is limited evidence regarding the effects of exergaming in pediatric-onset multiple sclerosis, especially in Türkiye. This single-center, randomized controlled trial aims to compare the effects of structured functional exercise training and exergaming-based rehabilitation in children and adolescents with POMS. The trial will evaluate physical activity levels, balance, fatigue, and quality of life. A total of 30 participants aged 12-22 years, diagnosed according to the revised 2017 McDonald criteria, and with an Expanded Disability Status Scale (EDSS) score below 6, will be randomly assigned to one of two groups. The conventional physiotherapy group will receive structured exercise training delivered through live Zoom sessions (tele-rehabilitation model). The exergaming group will perform interactive game-based exercises using the Nintendo Switch Ring Fit Adventure™ platform. Both interventions will run for 8 weeks, with sessions twice per week, each lasting 45 minutes, supervised by a physiotherapist. The Structured Functional Exercise Group will perform aerobic, strengthening, coordination, and balance exercises. The Exergaming Group will perform similar exercise components integrated into game scenarios. These scenarios provide visual and auditory feedback and motivation. Outcome assessments will be conducted before and after the intervention period. Assessments will include the following validated instruments: Physical activity level (Godin Leisure-Time Exercise Questionnaire and pedometer step count); Functional mobility (Six-Minute Walk Test and Timed Up and Go Test); Balance (Mini-BESTest Balance Scale); Fatigue (Pediatric Quality of Life Inventory - Multidimensional Fatigue Scale, PedsQL-MFS); Quality of life (Pediatric Quality of Life Inventory, PedsQL 4.0); Functional composite (Multiple Sclerosis Functional Composite, MSFC); and Lower limb strength (Five Times Sit-to-Stand Test). It is hypothesized that the exergaming program will produce improvements in physical activity levels, balance, fatigue perception, and quality of life compared to conventional exercise training. This study aims to provide evidence for the integration of technology-supported rehabilitation approaches into pediatric physiotherapy. It also aims to promote sustainable, motivating, and child-centered exercise models for POMS patients.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 12-22 years.
* Diagnosed with pediatric-onset multiple sclerosisaccording to the 2017 revised McDonald criteria.
* Expanded Disability Status Scale (EDSS) ≤ 6
* Participate in online exercise sessions via Zoom

Exclusion Criteria:

* Presence of orthopedic problems affecting mobility.
* Blurred vision or visual disturbances that could interfere with exergaming or exercise performance.
* Any comorbid medical, neurological, or psychiatric condition that could influence physical performance or study outcomes.
* History of relapse or corticosteroid treatment within the last three months.

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) | Baseline and at 8 weeks
  Time to rise from a chair, walk 3 m, turn, return, and sit. Shorter times indicate better mobility. It is an objective test used to assess functional mobility and balance in people with MS. Before the assessment, the patient is shown how the test will be performed. The patient is then asked to get up from a chair, walk 3 meters at a comfortable pace, and return to the chair and sit down. The test is repeated three times. The time taken in each attempt is recorded in seconds using a stopwatch.

SECONDARY OUTCOMES:
Mini-BESTest | Baseline and at 8 weeks
  The Mini-BESTest consists of 14 items or activities grouped into 4 sections: expected postural control (sitting to standing, toe-standing, standing on one leg), reactive postural control (compensatory stepping forward, backward, and sideways), sensory orientation (standing with eyes open on a firm surface, standing with eyes closed on a foam surface, standing with eyes closed on an inclined ramp), and dynamic gait (changing walking speed, walking with head turns, walking with pivot turns, stepping over an obstacle, timed stand and go with a dual task). The quality of performance on an item is represented by specific item scores (normal = 2, moderate = 1, and severe = 0) that add up to a total score ranging from 0 to 28. The expected postural control, reactive postural control, and sensory orientation section scores each range from 0 to 6, while the dynamic walking section score ranges from 0 to 10. Higher total and section scores indicate better balance control.
6 Minute Walk Test (6MWT) | Baseline and at 8 weeks
  It is a simple, practical test applied according to the standard protocol of the American Thoracic Society to measure walking capacity. It has been reported that the test is valid and reliable in MS patients with mild and moderate disability. In our study, 6 MWTs will be performed in accordance with the standards set in the guidelines for MS patients. The participant will be asked to walk as fast as possible at his own walking pace on the 30-meter track for 6 minutes. Before starting the test, participants will be explained that they can rest if they develop excessive fatigue or respiratory distress during the test and that this time is included in the test period. As a result of the test, the distance traveled by the participant will be recorded in meters.
Five Times Sit-to-Stand (5xSTS) | Baseline and at 8 weeks
  The arms are placed crosswise at chest level, and the patient is asked to sit down and stand up 5 times as quickly as possible from a standard chair. The test begins in a sitting position and ends in a sitting position. The result is recorded in seconds. This method, which is valid and reliable in MS, has been shown to be related to lower extremity muscle strength and balance. Lower times indicate higher performance. It is reliable in assessing lower extremity function.
Pedometer (Omron HJ-321-E) | Baseline and at 8 weeks
  It is an objective device used to assess physical activity levels and record the number of steps taken. Participants in the study will be provided with the Omron HJ-321-E brand pedometer, which is lightweight and easy to carry. All pedometers are calibrated with personalized measurements (step length, weight, height). Patients are asked to attach the pedometer to their non-dominant leg, either on a belt or clothing. The number of steps taken by participants over the course of one week will be recorded.
Godin Leisure-Time Exercise Questionnaire (GLTEQ) | Baseline and at 8 weeks
  This two-question survey measures individuals' physical activity behavior. The GBZEA is a simple, valid, and effective primary outcome measure for defining activity levels and tracking changes after an intervention. The first question asks how often light, moderate, and vigorous activities lasting over 15 minutes are performed in a typical week. The second asks how often activities causing sweating occur. To calculate the score, weekly frequencies are multiplied by 3, 5, and 9 metabolic equivalents (METs) for light, moderate, and vigorous activity, respectively. The moderate + vigorous score is obtained by adding moderate and vigorous points, while the total score is the sum of light, moderate, and vigorous activity points.
Multiple Sclerosis Functional Composite (MSFC) | Baseline and at 8 weeks
  It provides a more quantitative assessment than the EDSS. The Timed 25-Foot Walk (T25W) evaluates lower limb function by measuring the time needed to walk 8 meters (25 feet); it is repeated twice and averaged. The Nine Hole Peg Test (NHPT) measures upper limb function by timing how fast pegs are placed into nine holes; it is repeated twice for each hand and averaged. Cognitive function is assessed with the 3-second Paced Auditory Serial Addition Test (PASAT-3), where patients add each new number they hear to the previous one during a 3-minute test with 60 responses. The MSFC score combines results from all three tests into a single composite score using calculated z-scores.
Pediatric Quality of Life Multidimensional Fatigue Scale (PedsQL-MFS) | Baseline and at 8 weeks
  PedsQL-MFS total score (0-100 transformed).This scale is a valid and reliable measure for assessing fatigue levels in the pediatric population. It consists of two separate forms: self-report and proxy report. The versions for the 13-18 and 18-25 age groups will be used in this study. The 18-item symptom-focused scale assesses three areas of fatigue (general, sleep/rest, and cognitive). Items are reverse-scored, rated, and converted linearly to a 0-100 scale: 0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0. Higher scores indicate higher levels of fatigue. Higher scores represent less fatigue.
Pediatric Quality of Life Inventory (PedsQL) | Baseline and at 8 weeks
  It includes two parallel forms for children and families to complete and consists of sections on physical functions (8 items), emotional functions (5 items), social functions (5 items), and school functions (5 items). The child form has been developed for the 5-7, 8-12, 13-18, and 18-25 age groups, while the family form has been developed for the 2-4, 5-7, 8-12, 13-18, and 18-25 age groups. The inventory, prepared according to a five-point Likert scale, indicates that 0 = never caused a problem, 1 = hardly ever caused a problem, 2 = sometimes caused a problem, 3 = often caused a problem, and 4 = always caused a problem. A linear conversion is applied in calculating the total score of the scale, and the evaluation is made on a scale of 0-100 points (0=100, 1=75, 2=50, 3=25, 4=0). A high PedsQL score indicates better health-related quality of life. In our study, both the child and parent versions of the PedsQL will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Serhat Güler, Assoc. Prof., Study Chair — Istanbul University-Cerrahpasa Cerrahpasa Faculty of Medicine Department of Pediatric Neurology; Sema Saltık, Prof. Dr., Study Chair — Istanbul University-Cerrahpasa Cerrahpasa Faculty of Medicine, Department of Pediatric Neurology

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (including age, sex, and outcome measures) may be shared upon reasonable request, following approval by the ethics committee and the supervising institution.

REFERENCES:
- [Background] Sebastiao E, Sandroff BM, Learmonth YC, Motl RW. Validity of the Timed Up and Go Test as a Measure of Functional Mobility in Persons With Multiple Sclerosis. Arch Phys Med Rehabil. 2016 Jul;97(7):1072-7. doi: 10.1016/j.apmr.2015.12.031. Epub 2016 Mar 2. PMID 26944709
- [Background] Boiko A, Vorobeychik G, Paty D, Devonshire V, Sadovnick D; University of British Columbia MS Clinic Neurologists. Early onset multiple sclerosis: a longitudinal study. Neurology. 2002 Oct 8;59(7):1006-10. doi: 10.1212/wnl.59.7.1006. PMID 12370453
- [Background] Grover SA, Sawicki CP, Kinnett-Hopkins D, Finlayson M, Schneiderman JE, Banwell B, Till C, Motl RW, Yeh EA. Physical Activity and Its Correlates in Youth with Multiple Sclerosis. J Pediatr. 2016 Dec;179:197-203.e2. doi: 10.1016/j.jpeds.2016.08.104. Epub 2016 Oct 4. PMID 27717498
- [Background] Weikert M, Motl RW, Suh Y, McAuley E, Wynn D. Accelerometry in persons with multiple sclerosis: measurement of physical activity or walking mobility? J Neurol Sci. 2010 Mar 15;290(1-2):6-11. doi: 10.1016/j.jns.2009.12.021. Epub 2010 Jan 8. PMID 20060544
- [Background] Yeh EA, Kinnett-Hopkins D, Grover SA, Motl RW. Physical activity and pediatric multiple sclerosis: Developing a research agenda. Mult Scler. 2015 Nov;21(13):1618-25. doi: 10.1177/1352458515606526. Epub 2015 Oct 7. PMID 26447061
- [Background] Moller AB, Bibby BM, Skjerbaek AG, Jensen E, Sorensen H, Stenager E, Dalgas U. Validity and variability of the 5-repetition sit-to-stand test in patients with multiple sclerosis. Disabil Rehabil. 2012;34(26):2251-8. doi: 10.3109/09638288.2012.683479. Epub 2012 May 22. PMID 22612360
- [Background] Chan WLS, Chan CWL, Chan HHW, Chan KCK, Chan JSK, Chan OLW. A randomised controlled pilot study of a Nintendo Ring Fit Adventure balance and strengthening exercise program in community-dwelling older adults with a history of falls. Australas J Ageing. 2024 Sep;43(3):533-544. doi: 10.1111/ajag.13297. Epub 2024 Feb 26. PMID 38404233
- [Background] Alba-Rueda A, Lucena-Anton D, De Miguel-Rubio A. Effectiveness of two different exergaming systems in addition to conventional treatment for physical therapy in patients with multiple sclerosis: A study protocol for a multicenter, assessor-blind, 24-week, randomized controlled trial. Digit Health. 2024 Oct 18;10:20552076241287874. doi: 10.1177/20552076241287874. eCollection 2024 Jan-Dec. PMID 39430704
- [Background] Grover SA, Aubert-Broche B, Fetco D, Collins DL, Arnold DL, Finlayson M, Banwell BL, Motl RW, Yeh EA. Lower physical activity is associated with higher disease burden in pediatric multiple sclerosis. Neurology. 2015 Nov 10;85(19):1663-9. doi: 10.1212/WNL.0000000000001939. Epub 2015 Aug 12. PMID 26268901
- [Background] Polizzi A, Rinella S, Ruggieri M, Gentile AE, Verrelli CM, Iosa M. Efficacy of videogames and exergames in pediatric neurorehabilitation: a systematic review. Minerva Pediatr (Torino). 2024 Oct;76(5):690-702. doi: 10.23736/S2724-5276.23.07146-X. Epub 2023 Jun 16. PMID 37335184
- [Background] Sikes EM, Richardson EV, Motl RW. A Qualitative Study of Exercise and Physical Activity in Adolescents with Pediatric-Onset Multiple Sclerosis. Int J MS Care. 2019 Mar-Apr;21(2):81-91. doi: 10.7224/1537-2073.2018-033. PMID 31049039
- [Background] Yazgan YZ, Tarakci E, Tarakci D, Ozdincler AR, Kurtuncu M. Comparison of the effects of two different exergaming systems on balance, functionality, fatigue, and quality of life in people with multiple sclerosis: A randomized controlled trial. Mult Scler Relat Disord. 2020 Apr;39:101902. doi: 10.1016/j.msard.2019.101902. Epub 2019 Dec 21. PMID 31924591
- [Background] Vural P, Zenginler Yazgan Y, Tarakci E, Guler S, Saltik S. The effects of online exercise training on physical functions and quality of life in patients with pediatric-onset multiple sclerosis. Mult Scler Relat Disord. 2023 Jun;74:104710. doi: 10.1016/j.msard.2023.104710. Epub 2023 Apr 9. PMID 37086635